CLINICAL TRIAL: NCT05652049
Title: An Exploratory Study Using New Ultrasound Techniques to Assess Peritoneal Fibrosis and Encapsulating Peritoneal Sclerosis in Peritoneal Dialysis Patients
Brief Title: Using New Ultrasound Techniques to Assess Peritoneal Fibrosis in Peritoneal Dialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Na Jiang, Associate Chief Physician of Nephrology, Shanghai Jiao Tong University School of Medicine
Other Study IDs: new ultrasound technology
Record Dates: First submitted 2022-12-08; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Peritoneal Sclerosis
MeSH Terms: conditions — Peritoneal Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- short-term peritoneal dialysis: the time of treatment of peritoneal dialysis less 12 months
- long-term peritoneal dialysis: the time of treatment of peritoneal dialysis more than 10 years

SUMMARY:
Explore the role of new ultrasound techniques in the assessment of peritoneal fibrosis and encapsulating peritoneal sclerosis in peritoneal dialysis patients

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients on PD
* PD duration ≤12 months or ≥10 years
* Age between 18-75years

Exclusion Criteria:

* Refusing to sign up informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage renal diseases（ESRD） patients on PD
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
parietal peritoneal fibrosis | the 1 day when being recruited
  Ultrasonography evaluates parietal peritoneal fibrosis, including parameters such as thickness, stiffness, elasticity, and blood supply.

SECONDARY OUTCOMES:
encapsulting peritoneal sclerosis | the 1 day when being recruited
  Ultrasonography assesses for encapsulting peritoneal sclerosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No